CLINICAL TRIAL: NCT01629784
Title: Effectiveness of a Knowledge-based Intervention for Patients With Cutaneous Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Assistant Professor of Dermatology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: STU65095
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-04

CONDITIONS: Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CLE and sun counseling (Other)
  Interventions: Behavioral: Cutaneous Lupus educational script

INTERVENTIONS:
Behavioral: Cutaneous Lupus educational script — Subjects will listen to a short informational script on Cutaneous lupus and skin protection

SUMMARY:
Studies have shown that there are significant differences in severity and outcome of lupus in patients of colored skin compared with Caucasians. There are many factors that lead to this discrepancy: genetics, poverty, education level, as well as behavioral and cultural factors. Cutaneous Lupus Erythematosus (CLE) is a disease of flares and remissions with identifiable triggers. One of the most aggravating triggers in CLE is sun exposure. The investigators hypothesize that there are disparities in knowledge about photoprotection, leading to poorer outcomes in minority ethnic groups. This study aims to assess knowledge of risk factors and triggers, especially sun exposure, and the effects on quality of life of Caucasian and minority populations, by conducting an assessment survey and subsequent teaching intervention on appropriate skin protection techniques including appropriate sun screen application, and use of sun-protective clothing. After three months a survey to evaluate knowledge retention about and the application of the educational intervention will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of cutaneous lupus erythematous
* Subjects ages 18 years of age and older and able to give consent

Exclusion Criteria:

* That which does not fit the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Kundu, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Finlay AY. Quality of life assessments in dermatology. Semin Cutan Med Surg. 1998 Dec;17(4):291-6. doi: 10.1016/s1085-5629(98)80026-6. PMID 9859917
- [Background] Foering K, Goreshi R, Klein R, Okawa J, Rose M, Cucchiara A, Werth VP. Prevalence of self-report photosensitivity in cutaneous lupus erythematosus. J Am Acad Dermatol. 2012 Feb;66(2):220-8. doi: 10.1016/j.jaad.2010.12.006. Epub 2011 Jul 13. PMID 21742409
- [Background] Kundu RV, Kamaria M, Ortiz S, West DP, Rademaker AW, Robinson JK. Effectiveness of a knowledge-based intervention for melanoma among those with ethnic skin. J Am Acad Dermatol. 2010 May;62(5):777-84. doi: 10.1016/j.jaad.2009.08.047. Epub 2010 Mar 9. PMID 20219266
- [Background] Werth VP. Clinical manifestations of cutaneous lupus erythematosus. Autoimmun Rev. 2005 Jun;4(5):296-302. doi: 10.1016/j.autrev.2005.01.003. Epub 2005 Feb 10. PMID 15990077
- See also: Northwestern University Department of Dermatology Actively Enrolling Research Trials — http://www.feinberg.northwestern.edu/depts/dermatology/research/clinical-trials/ctu-active%20trials.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult subjects with cutaneous lupus erythematosus (CLE) were recruited from Northwestern University's dermatology and rheumatology clinics.
Groups:
- Cutaneous Lupus Erythematosus (CLE): Subjects completed a written questionnaire to collect demographic data, including personal history of CLE and sun protection behaviors, and to assess knowledge about CLE and sun protection. Next, subjects listened to a scripted, educational lecture about CLE and sun protection, and then immediately completed a post-lecture written questionnaire to assess knowledge about CLE and sun protection. Three months after the educational lecture, subjects were contacted by phone to complete a final knowledge and behavioral assessment.
Period: Overall Study
Arm/Group | Cutaneous Lupus Erythematosus (CLE)
Started | 31
Completed | 25
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Cutaneous Lupus Erythematosus (CLE)
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Correctly Answered a Knowledge Assessment Item Immediately Before and After an Educational Lecture
Description: In order to evaluate the immediate effect of an educational lecture about cutaneous lupus erythematosus (CLE) and sun protection, subjects completed a written questionnaire to assess knowledge about CLE and sun protection immediately before and after the educational lecture. The percentage of subjects who correctly answered a knowledge assessment item were calculated pre- and post-educational lecture.
Time Frame: immediately before and after an educational lecture
Measure: Number; unit: percentage of participants
Groups:
- Pre-educational Lecture; Post-educational Lecture: Subjects completed a written questionnaire to collect demographic data, including personal history of CLE and sun protection behaviors, and to assess knowledge about CLE and sun protection. Next, subjects listened to a scripted, educational lecture about CLE and sun protection, and then immediately completed a written questionnaire to assess knowledge about CLE and sun protection.
Arm/Group | Pre-educational Lecture | Post-educational Lecture
Number analyzed (Participants) | 31 | 31
percentage of participants
  Risk of lupus for people of color | 52 | 94
  Smoking linked to lupus | 19 | 90
  Sun exposure linked to lupus | 81 | 97
  Sun brings out lupus lesions | 74 | 97
  Should use sun-protective clothing to protect skin | 94 | 100
  Should apply sunscreen before going outdoors | 97 | 100
  Time to apply sunscreen before sun exposure | 39 | 48
  Type of sunscreen that should be used | 87 | 90
  Exposure to UV rays while indoors through glass | 68 | 100
  Exposure to UV rays with indoor tanning | 39 | 100
  Should apply sunscreen under makeup | 68 | 100
  Should avoid sun during hours of 10 am - 2 pm | 84 | 100

2. Secondary Outcome: Percentage of Subjects Who Correctly Answered a Knowledge or Behavioral Assessment Item Before and 3 Months After an Educational Lecture
Description: In order to evaluate the long-term effect of an educational lecture about cutaneous lupus erythematosus (CLE) and sun protection, subjects completed a questionnaire to assess knowledge about CLE and sun protection behaviors immediately before and three months after an educational lecture. The percentage of subjects who correctly answered a knowledge or behavioral assessment item were calculated pre- and three months post-educational lecture.
Time Frame: before and 3 months after an educational lecture
Measure: Number; unit: percentage of participants
Groups:
- Pre-educational Lecture; Three Months Post-educational Lecture: Subjects completed a written questionnaire to collect demographic data, including personal history of CLE and sun protection behaviors, and to assess knowledge about CLE and sun protection. Next, subjects listened to a scripted, educational lecture about CLE and sun protection. 3 months later, subjects were contacted by phone to complete a knowledge and behavioral assessment about CLE and sun protection.
Arm/Group | Pre-educational Lecture | Three Months Post-educational Lecture
Number analyzed (Participants) | 31 | 25
percentage of participants
  Smoking linked to lupus | 19 | 45
  Sun exposure linked to lupus | 81 | 77
  Sun brings out lupus lesions | 74 | 77
  Should use sun-protective clothing to protect skin | 94 | 71
  Seek medical care for change in rash appearance | 97 | 81
  Apply sunscreen before going outdoors | 71 | 71
  Apply sunscreen at correct time prior to exposure | 32 | 45
  Apply correct type of sunscreen | 58 | 58
  Reapply sunscreen at correct time if dry | 19 | 13
  Reapply sunscreen at correct time if wet | 23 | 19
  Avoid more than two hours of sun exposure | 25 | 26
  Limit outdoor social gatherings | 55 | 48
  Wear sun-protective clothing | 68 | 81
  Avoid indoor tanning | 94 | 81
  Apply sunscreen under makeup | 45 | 52
  Avoid sun exposure between 10 am - 2 pm | 71 | 71

ADVERSE EVENTS:
Arm/Group | Cutaneous Lupus Erythematosus (CLE)
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes